CLINICAL TRIAL: NCT02264626
Title: Effects of Remifentanil Based Sedation on Patient-ventilator Interaction, in Patients Undergoing Noninvasive Ventilation (NIV)
Brief Title: Sedation During Noninvasive Ventilation (NIV)
Acronym: REMI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, dr. Stefano Nava, Professor of Respiratory Medicine, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 116/2014O
Record Dates: First submitted 2014-10-04; First posted 2014-10-15 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-10

CONDITIONS: Acute Hypercapnic Respiratory Failure
Keywords: acute respiratory failure; noninvasive ventilation; sedation; patient/ventilator interaction
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Remifentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- acutely ill patients (Experimental): administration of remifentanil at the infusion rate by 0.025 μg kg-1 min-1 to a maximum of 0.10 μg kg-1 min-1.
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Remifentanil — infusion at a rate by 0.025 μg kg-1 min-1 every minute to a maximum of 0.15 μg kg-1 min-1.
  Other Names: ultriva

SUMMARY:
In patients undergoing NIV for acute respiratory, lack of tolerance is one of the main reason of failure.

This may result in a poor synchrony between the patient and the machine, leading to gross mismatching and potentially to an increased work of breathing.

The investigators aim to investigate whether in these patients poorly responding to NIV the use of a sedation protocol using remifentanil will lead to an improve patient-ventilator interaction and better compliance to NIV.

DETAILED DESCRIPTION:
In patients undergoing NIV for acute respiratory, lack of tolerance is one of the main reason of failure.

This may result in a poor synchrony between the patient and the machine, leading to gross mismatching and potentially to an increased work of breathing.

The investigators aim to investigate whether in these patients poorly responding to NIV the use of a sedation protocol using remifentanil will lead to an improve patient-ventilator interaction and better compliance to NIV.

In this physiological study the investigators will study 15 patients at risk of failing NIV because of scarce tolerance and showing clinical signs of poor interaction with the ventilator.

Once the patient will be enrolled the investigators will record using the balloon-catheter technique the online measurement of respiratory mechanics, to assess the inspiratory muscle effort and the matching between the patient breathing pattern and that of the ventilator The investigators will also record the clinical success of sedation (i.e. need or not for endotracheal intubation)

ELIGIBILITY:
Inclusion Criteria:

* Ph<7,35 and PaCO2>50 mmHg with acute respiratory failure
* Signs of respiratory distress and poor synchrony with the ventilator as assessed on the ventilator screen and by looking patient own rate and ventilator recorded rate

Exclusion Criteria:

* Patients responding well to NIV and not showing signs of poor synchrony

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2014-10; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
patient-ventilator interaction | one hour
  patient-ventilator interaction will be assessed using the recording of respiratory mechanics to identify
matching of inspiratory timing | one hour
  the patients inspiratory time vs ventilator inspiratory time
Wasted efforts | one hour
  breaths unable to trigger the ventilator

SECONDARY OUTCOMES:
NIV failure | one hour
  failure will be defined as the need for intubation:
  * gasping for air
  * worsening of sensorium
  * respiratory arrest
  * retention of secretions and/ or death

CONTACTS AND LOCATIONS:
Overall Officials: stefano nava, md, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- San'Orsola Malpighi Hospital, Bologna ITALY, Bologna, Italy